CLINICAL TRIAL: NCT00773643
Title: Osteogenic Profiling of Tissue From Children With Craniosynostosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Joseph Losee, Ross H. Musgrave Professor of Pediatric Plastic Surgery Executive Vice-Chair and Program Director Department of Plastic Surgery University of Pittsburgh Medical Center, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07110284
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Craniosynostosis
Keywords: to procure human temporalis muscle, subcutaneous adipose (fat), and bone tissue samples from children with craniosynostosis,; to grow cells from these tissues in vitro; to evaluate the osteogenic potentials of these cell types.
MeSH Terms: conditions — Craniosynostoses; Platelet Glycoprotein IV Deficiency | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tissue Sample (Experimental): A biopsy of the patient's temporalis muscle, subcutaneous adipose, and bone tissue is the experimental procedure. The procedure will not involve any extra incisions or dissection, as these tissues will be exposed during the reconstructive procedure. A very small fragment of each tissue type, 2mm X 2mm X 3mm biopsy, will be removed.
  Interventions: Other: biopsy

INTERVENTIONS:
Other: biopsy — A biopsy of the patient's temporalis muscle, subcutaneous adipose, and bone tissue is the experimental procedure. The procedure will not involve any extra incisions or dissection, as these tissues will be exposed during the reconstructive procedure. A very small fragment of each tissue type, 2mm X 2mm X 3mm biopsy, will be removed.

SUMMARY:
The primary objectives of this study are

* to procure human temporalis muscle, subcutaneous adipose (fat), and bone tissue samples from children with craniosynostosis,
* to grow cells from these tissues in vitro,
* to evaluate the osteogenic potentials of these cell types.

DETAILED DESCRIPTION:
The screening procedures include review and collection of information from the patient's medical record, Name, Date of Birth, Medical record number, clinical diagnosis of classification of craniosynostosis, genetic screen for syndromic synostosis (FGFR, TWIST, MSX2 mutation screen), and a clinical examination at the Cleft -Craniofacial Center. During the clinical examination, the plastic surgeon will determine the presence of a craniosynostosis and the need for surgical intervention. The evaluation and surgical repair of these patients with craniosynostosis will not differ from normal, nor from the current standard of care.

In order to reconstruct, reshape, and expand the contours of the deformed craniofacial skeleton, large skin incisions and subcutaneous dissections are necessary to allow for sufficient exposure during the procedure. These large incisions and dissections are a necessary part of the reconstruction. During the normal course of the procedure, temporalis muscle, a muscle of mastication in the temporal area, and subcutaneous adipose will be visible and exposed. It is only after the plastic surgeon has obtained this standard exposure that excisional biopsies of a maximum size of 2mm X 2mm X 3mm will be taken from consented patients. Bone samples will be collected from bone tissue that would normally be discarded during the reconstructive surgery, so no additional procedures are needed to collect the bone samples. Biopsy samples will not be provided to secondary investigators. The muscle and adipose biopsies are research required procedures. At the time of surgery one sample of tissue will be taken from temporalis muscle, subcutaneous adipose, and bone. The investigator will review the results of the test/procedure that are part of the standard of care and results will become part of the research record. The investigators will continue to use and disclose identifiable medical information and keep stored tissue samples for seven years. After this seven year period, all identifying information will be removed samples will be destroyed.

The muscle and adipose tissue biopsies will take approximately 10 minutes. The samples of bone tissue will be discarded as a result of the reconstructive surgery and will, therefore, not add any time to the surgical procedure.

Subjects will not be notified of the results of this study because the results will not impact the clinical care of the subject.

ELIGIBILITY:
Inclusion Criteria:

* Children with craniosynostosis undergoing surgical calvarial reconstruction between the ages of 2 months of age to 18 years old will be included in this study. This surgery is the standard of care in the sequence of treatment for craniosynostosis patients. Pediatric plastic surgeons at the Cleft-Craniofacial Center at Children's Hospital of Pittsburgh of UPMC work primarily with children as part of their patient populations and are trained for this during their residencies. Children will be evaluated initially at the Pittsburgh Cleft Palate and Craniofacial Center at Children's Hospital of Pittsburgh which is set up to accommodate children of all ages and their families.
* Approximately twelve to twenty children are normally treated in this facility each year.
* All patients will be asked to contribute to this study.
* The research study satisfies risk Criterion 3 (45 CFR 46.406) for the inclusion of children in research whereas the research involves an intervention or procedure that presents greater than minimal risk to the involved children and which does not hold out the potential for direct individual benefit. Pediatric patients undergoing surgical repair craniosynostosis normally do not have a biopsy of the temporalis muscle or the adipose tissue of the scalp (experimental procedures). These biopsies will be performed by a plastic surgeon who is experienced in the surgical repair of pediatric patients and poses no additional likely or common risks above the surgical repair of the calvaria. Infrequent risks may include a slight increase in bleeding representing a few more drops of blood loss. Rare risks, occurring in less than one percent of patients, may subject the patient to injury to nerves in a small area of the biopsy which may result in a decrease of muscle function in that area. This intervention could provide detailed, basic information regarding the relationship between the progenitor cells and craniosynostosis.

Exclusion Criteria:

* All patients not undergoing calvarial reconstruction to correct craniosynostosis will be excluded from this study.
* Selection will be based on an individual's willingness to participate in the study.
* A subject will also be removed from the research study if the targeted muscle, adipose, or bone tissues are unavailable due to necrosis, infection, or if the removal of the tissues may adversely effect the surgical outcome in some way.

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
The investigators will attempt to correlate patient diagnosis with a cellular biological response. Similar work has not yet been performed, making this study a pilot study based on such a correlation. | 2 years or 50 subject, Which ever happens first

CONTACTS AND LOCATIONS:
Overall Officials: Jospeh Losee, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Joseph Losee, MD, Pittsburgh, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania